CLINICAL TRIAL: NCT05597709
Title: Prevalence of Metabolic Associated Fatty Liver Disease in Patients With Type 2 Diabetes in Jiangsu Province of China: a Prospective, Multicenter, Real-world Study
Brief Title: Prevalence of MAFLD in Patients With Type 2 Diabetes in Jiangsu Province of China
Status: Recruiting | Type: Observational
Sponsor: Wuxi Hisky Medical Technology Co Ltd (Industry)
Collaborators: Zhongda Hospital (Other); Suzhou Municipal Hospital (Other); Suzhou Fifth People's Hospital (Unknown); Xuzhou Mining Group General Hospital (Unknown); Nantong First People's Hospital (Other); Changzhou Second People's Hospital (Unknown); Huaian Second People's Hospital (Unknown); Huaian Hospital (Unknown); Taizhou Jiangyan Traditional Chinese Medicine Hospital (Unknown); Yangzhou Jiangdu People's Hospital (Unknown); Huaian Xuyi County People's Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: MAFLD
Record Dates: First submitted 2022-10-24; First posted 2022-10-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Type 2 Diabetes Mellitus in Remission; Metabolic Associated Fatty Liver Disease
Keywords: Type 2 diabetes mellitus; Metabolic associated fatty liver disease; ultrasound attenuation parameter
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biospecimen including blood samples for blood glucose measurement (fasting blood glucose, glycosylated hemoglobin), fasting insulin level, biochemical examination (PLT, AST, ALT, ALP, GGT, TBIL, DBIL, TC, TG, LDL-C, HDL-C, etc.), and FIB-4(PC III, IV-C, LN, HA）.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who diagnosed as T2DM: Diagnosed as T2DM according to the Chinese Guidelines for the Prevention and Treatment of Type 2 Diabetes
  Interventions: Procedure: Ultrasound attenuation parameter measurement, fasting blood glucose and fasting insulin determination

INTERVENTIONS:
Procedure: Ultrasound attenuation parameter measurement, fasting blood glucose and fasting insulin determination — Eligible participants will receive ultrasound attenuation parameter with iLivTouch, fasting blood glucose and fasting insulin determination

SUMMARY:
In 2019, the number of patients with diabetes was about 463 million in the world, accounting for 8.3% of the total population, and it is expected to rise to 578 million (9.2%) by 2030 and 700 million (9.6%) by 2045. According to the WHO diagnostic criteria, the prevalence of diabetes among adults in China from 2015 to 2017 was 11.2%, of which over 90% were type 2 diabetes mellitus (T2DM). The global prevalence of non-alcoholic fatty liver disease (NAFLD) is also very high, which was approximately 25% in 2016. The prevalence of NAFLD may continue to rise. NAFLD is often accompanied by clinical manifestations of metabolic syndrome, such as obesity, T2DM, hyperlipidemia and hypertension.

DETAILED DESCRIPTION:
The presence of NAFLD not only increases the risk of T2DM, but also accelerates the process of various diabetes-related organ damage in patients with T2DM. Similarly, T2DM also increases the risk of NAFLD. However, in patients with T2DM, there are few reports on the correlation between ultrasound attenuation parameters for non-invasive assessment of liver fat content and insulin resistance. In addition, T2DM may be the most important predictor of adverse clinical outcomes in NAFLD patients. T2DM is an important predictor of NAFLD patients progressing to compensated advanced chronic liver disease (cACLD), and even cirrhotic portal hypertension and other end-stage liver diseases.

In February 2020, international experts suggested NAFLD to be renamed metabolic associated fatty liver disease (MAFLD). In April of the same year, the Journal of Hepatology released a new definition and diagnosis of MAFLD with the criteria based on histological (liver biopsy), imaging, or blood biomarker indicating the presence of hepatic fat accumulation (hepatocyte steatosis), in combination with one of the following 3 conditions: overweight/obesity, type 2 diabetes and metabolic dysfunction. The new diagnostic criteria are based on underlying metabolic abnormalities and recognize that MAFLD often coexists with other diseases.

Therefore, this study aims to investigate the prevalence and clinical characteristics of MAFLD in patients with T2DM, as well as the correlation between UAP and insulin resistance in T2DM. Patients will be followed up to 5 years for the clinical outcomes at 3months, 6 months, 12 months, 36 months, 48 months and 60 months respectively and the risk factors affecting the clinical outcomes of patients with T2DM will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as T2DM according to the Chinese Guidelines for the Prevention and Treatment of Type 2 Diabetes
* UAP were measured based on iLivTouch
* Willing to attend this study and able to provide the written informed consent.

Exclusion Criteria:

* Other types of diabetes
* Patients unable to receive regular follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with T2DM
Sampling Method: Probability Sample
Enrollment: 2900 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with MAFLD in the T2DM population screened by UAP with iLivTouch | 12 months
  To explore the prevalence and clinical characteristics of MAFLD in patients with T2DM
Correlation between UAP and insulin resistance | 12 months
  To explore the correlation between UAP and insulin resistance in patients with T2DM
Analysis of risk factors for clinical outcomes in patients with T2DM | 5 years
  To analyze risk factors affecting clinical outcomes in patients with T2DM

CONTACTS AND LOCATIONS:
Overall Officials: Ling Li, Professor, Principal Investigator — Zhongda Hospital
Locations (1):
- Zhongda Hospital, Medical School, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saeedi P, Petersohn I, Salpea P, Malanda B, Karuranga S, Unwin N, Colagiuri S, Guariguata L, Motala AA, Ogurtsova K, Shaw JE, Bright D, Williams R; IDF Diabetes Atlas Committee. Global and regional diabetes prevalence estimates for 2019 and projections for 2030 and 2045: Results from the International Diabetes Federation Diabetes Atlas, 9th edition. Diabetes Res Clin Pract. 2019 Nov;157:107843. doi: 10.1016/j.diabres.2019.107843. Epub 2019 Sep 10. PMID 31518657
- [Background] Chalasani N, Younossi Z, Lavine JE, Charlton M, Cusi K, Rinella M, Harrison SA, Brunt EM, Sanyal AJ. The diagnosis and management of nonalcoholic fatty liver disease: Practice guidance from the American Association for the Study of Liver Diseases. Hepatology. 2018 Jan;67(1):328-357. doi: 10.1002/hep.29367. Epub 2017 Sep 29. No abstract available. PMID 28714183
- [Background] Younossi ZM, Koenig AB, Abdelatif D, Fazel Y, Henry L, Wymer M. Global epidemiology of nonalcoholic fatty liver disease-Meta-analytic assessment of prevalence, incidence, and outcomes. Hepatology. 2016 Jul;64(1):73-84. doi: 10.1002/hep.28431. Epub 2016 Feb 22. PMID 26707365
- [Background] Byrne CD, Targher G. NAFLD: a multisystem disease. J Hepatol. 2015 Apr;62(1 Suppl):S47-64. doi: 10.1016/j.jhep.2014.12.012. PMID 25920090
- [Background] Younossi Z, Anstee QM, Marietti M, Hardy T, Henry L, Eslam M, George J, Bugianesi E. Global burden of NAFLD and NASH: trends, predictions, risk factors and prevention. Nat Rev Gastroenterol Hepatol. 2018 Jan;15(1):11-20. doi: 10.1038/nrgastro.2017.109. Epub 2017 Sep 20. PMID 28930295
- [Background] Lyu K, Zhang Y, Zhang D, Kahn M, Ter Horst KW, Rodrigues MRS, Gaspar RC, Hirabara SM, Luukkonen PK, Lee S, Bhanot S, Rinehart J, Blume N, Rasch MG, Serlie MJ, Bogan JS, Cline GW, Samuel VT, Shulman GI. A Membrane-Bound Diacylglycerol Species Induces PKCϵ-Mediated Hepatic Insulin Resistance. Cell Metab. 2020 Oct 6;32(4):654-664.e5. doi: 10.1016/j.cmet.2020.08.001. Epub 2020 Sep 2. PMID 32882164
- [Background] Hossain N, Afendy A, Stepanova M, Nader F, Srishord M, Rafiq N, Goodman Z, Younossi Z. Independent predictors of fibrosis in patients with nonalcoholic fatty liver disease. Clin Gastroenterol Hepatol. 2009 Nov;7(11):1224-9, 1229.e1-2. doi: 10.1016/j.cgh.2009.06.007. Epub 2009 Jun 25. PMID 19559819
- [Background] Stepanova M, Rafiq N, Makhlouf H, Agrawal R, Kaur I, Younoszai Z, McCullough A, Goodman Z, Younossi ZM. Predictors of all-cause mortality and liver-related mortality in patients with non-alcoholic fatty liver disease (NAFLD). Dig Dis Sci. 2013 Oct;58(10):3017-23. doi: 10.1007/s10620-013-2743-5. Epub 2013 Jun 18. PMID 23775317
- [Background] Fracanzani AL, Valenti L, Bugianesi E, Andreoletti M, Colli A, Vanni E, Bertelli C, Fatta E, Bignamini D, Marchesini G, Fargion S. Risk of severe liver disease in nonalcoholic fatty liver disease with normal aminotransferase levels: a role for insulin resistance and diabetes. Hepatology. 2008 Sep;48(3):792-8. doi: 10.1002/hep.22429. PMID 18752331
- [Background] Younossi ZM, Golabi P, de Avila L, Paik JM, Srishord M, Fukui N, Qiu Y, Burns L, Afendy A, Nader F. The global epidemiology of NAFLD and NASH in patients with type 2 diabetes: A systematic review and meta-analysis. J Hepatol. 2019 Oct;71(4):793-801. doi: 10.1016/j.jhep.2019.06.021. Epub 2019 Jul 4. PMID 31279902
- [Background] Baffy G, Brunt EM, Caldwell SH. Hepatocellular carcinoma in non-alcoholic fatty liver disease: an emerging menace. J Hepatol. 2012 Jun;56(6):1384-91. doi: 10.1016/j.jhep.2011.10.027. Epub 2012 Feb 9. PMID 22326465
- [Background] Rafiq N, Bai C, Fang Y, Srishord M, McCullough A, Gramlich T, Younossi ZM. Long-term follow-up of patients with nonalcoholic fatty liver. Clin Gastroenterol Hepatol. 2009 Feb;7(2):234-8. doi: 10.1016/j.cgh.2008.11.005. Epub 2008 Nov 7. PMID 19049831
- [Background] Stepanova M, Rafiq N, Younossi ZM. Components of metabolic syndrome are independent predictors of mortality in patients with chronic liver disease: a population-based study. Gut. 2010 Oct;59(10):1410-5. doi: 10.1136/gut.2010.213553. Epub 2010 Jul 26. PMID 20660697
- [Background] Qi X, Berzigotti A, Cardenas A, Sarin SK. Emerging non-invasive approaches for diagnosis and monitoring of portal hypertension. Lancet Gastroenterol Hepatol. 2018 Oct;3(10):708-719. doi: 10.1016/S2468-1253(18)30232-2. PMID 30215362
- [Background] Qu Y, Song YY, Chen CW, Fu QC, Shi JP, Xu Y, Xie Q, Yang YF, Zhou YJ, Li LP, Xu MY, Cai XB, Zhang QD, Yu H, Fan JG, Lu LG. Diagnostic Performance of FibroTouch Ultrasound Attenuation Parameter and Liver Stiffness Measurement in Assessing Hepatic Steatosis and Fibrosis in Patients With Nonalcoholic Fatty Liver Disease. Clin Transl Gastroenterol. 2021 Apr 13;12(4):e00323. doi: 10.14309/ctg.0000000000000323. PMID 33848277
- [Background] Duan WJ, Wang XZ, Ma AL, Shang J, Nan YM, Gao ZL, Tang H, Fu QC, Xie Q, Mao Q, Niu JQ, Han T, Li J, Han Y, Cao JB, Kong YY, Shi XY, Lv FD, Wang TL, Ma H, You H, Ou XJ, Jia JD. Multicenter prospective study to validate a new transient elastography device for staging liver fibrosis in patients with chronic hepatitis B. J Dig Dis. 2020 Sep;21(9):519-525. doi: 10.1111/1751-2980.12924. PMID 32700794
- [Background] Eslam M, Sanyal AJ, George J; International Consensus Panel. MAFLD: A Consensus-Driven Proposed Nomenclature for Metabolic Associated Fatty Liver Disease. Gastroenterology. 2020 May;158(7):1999-2014.e1. doi: 10.1053/j.gastro.2019.11.312. Epub 2020 Feb 8. PMID 32044314
- [Background] Eslam M, Newsome PN, Sarin SK, Anstee QM, Targher G, Romero-Gomez M, Zelber-Sagi S, Wai-Sun Wong V, Dufour JF, Schattenberg JM, Kawaguchi T, Arrese M, Valenti L, Shiha G, Tiribelli C, Yki-Jarvinen H, Fan JG, Gronbaek H, Yilmaz Y, Cortez-Pinto H, Oliveira CP, Bedossa P, Adams LA, Zheng MH, Fouad Y, Chan WK, Mendez-Sanchez N, Ahn SH, Castera L, Bugianesi E, Ratziu V, George J. A new definition for metabolic dysfunction-associated fatty liver disease: An international expert consensus statement. J Hepatol. 2020 Jul;73(1):202-209. doi: 10.1016/j.jhep.2020.03.039. Epub 2020 Apr 8. PMID 32278004
- [Background] de Franchis R; Baveno VI Faculty. Expanding consensus in portal hypertension: Report of the Baveno VI Consensus Workshop: Stratifying risk and individualizing care for portal hypertension. J Hepatol. 2015 Sep;63(3):743-52. doi: 10.1016/j.jhep.2015.05.022. Epub 2015 Jun 3. No abstract available. PMID 26047908
- [Background] Bhardwaj A, Kedarisetty CK, Vashishtha C, Bhadoria AS, Jindal A, Kumar G, Choudhary A, Shasthry SM, Maiwall R, Kumar M, Bhatia V, Sarin SK. Carvedilol delays the progression of small oesophageal varices in patients with cirrhosis: a randomised placebo-controlled trial. Gut. 2017 Oct;66(10):1838-1843. doi: 10.1136/gutjnl-2016-311735. Epub 2016 Jun 13. PMID 27298379
- [Background] Abraldes JG, Bureau C, Stefanescu H, Augustin S, Ney M, Blasco H, Procopet B, Bosch J, Genesca J, Berzigotti A; Anticipate Investigators. Noninvasive tools and risk of clinically significant portal hypertension and varices in compensated cirrhosis: The "Anticipate" study. Hepatology. 2016 Dec;64(6):2173-2184. doi: 10.1002/hep.28824. Epub 2016 Oct 27. PMID 27639071
- [Background] Chinese Diabetes Society. Guideline for the prevention and treatment of type 2 diabetes mellitus in China(2020 edition). Chinese Journal of Endocrinology and Metabolism. 2021;4:311-398.
- [Background] Chinese Society of Endocrinology;Chinese Diabetes Society;Zhu Dulong;Zhao Jiajun;Mu Yiming.Management of Chinese adults with type 2 diabetes and non-alcoholic fatty liver disease:an expert consensus.Chinese Journal of Endocrinology and Metabolism.2021;7:589-598.
- [Background] Lai SQ, Hong ZZ, Chen HM, Lin JX, Kuang J, Li YB. [Correlation between ectopic fat accumulation and insulin sensitivity in obese individuals with different glucose tolerance levels]. Nan Fang Yi Ke Da Xue Xue Bao. 2017 Nov 20;37(11):1461-1466. doi: 10.3969/j.issn.1673-4254.2017.11.06. Chinese. PMID 29180325
- [Background] Qi XL. [Cirrhotic portal hypertension in the non-invasive era: what we grasp]. Zhonghua Gan Zang Bing Za Zhi. 2018 Apr 20;26(4):241-244. doi: 10.3760/cma.j.issn.1007-3418.2018.04.001. Chinese. PMID 29996331
- [Background] XiaoYuan X etal.Guidelines for the diagnosis and treatment of esophageal and gastric variceal bleeding in cirrhotic portal hypertension.Journal of Clinical Hepatology.2016;2:203-219
- [Background] Zuo ZB, Cui HZ, Huang CX, Guo Y, Pan KR, Wang MC, Du W, Huang B, Xu AF. [Clinical study of FibroTouch and six serological models for assessing the degree of liver fibrosis in patients with chronic hepatitis B]. Zhonghua Gan Zang Bing Za Zhi. 2019 Jun 20;27(6):430-435. doi: 10.3760/cma.j.issn.1007-3418.2019.06.008. Chinese. PMID 31357758
- [Derived] Huang N, Su X, Yu T, Wu X, Lu B, Sun W, Yao L, Wang M, Wang Y, Wu W, Liu Y, Yang T, Gao R, Miao C, Li L. Serum 25-hydroxy vitamin D level is associated with elastography-detected liver fibrosis in patients with type 2 diabetes mellitus in China. Front Endocrinol (Lausanne). 2024 Nov 29;15:1420088. doi: 10.3389/fendo.2024.1420088. eCollection 2024. PMID 39698035
- [Derived] Yu H, Su X, Tao W, Sun W, Zhang X, Han Q, Zhao Z, Zhang Y, Chen X, Liu X, Jia D, Fang L, Li L. Prevalence and characteristics of liver steatosis and fibrosis in type 2 diabetes mellitus (T2DM) patients: a cross-sectional study in populations of eastern China. BMJ Open. 2024 Dec 12;14(12):e087550. doi: 10.1136/bmjopen-2024-087550. PMID 39672583